CLINICAL TRIAL: NCT03770364
Title: Peri-operative Hypothermia in Children: Improving Outcomes With Risk Prediction
Brief Title: Peri-operative Hypothermia in Children
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017/2298
Record Dates: First submitted 2017-08-27; First posted 2018-12-10 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-02

CONDITIONS: Hypothermia Following Anesthesia, Sequela; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the incidence of hypothermia in the local paediatric population in the peri-operative period, identify the risk factors involved, and thereafter develop and implement clinical practice guidelines to reduce IPH such that temperature monitoring and heat conservation measures can be implemented in a cost-effective way. The secondary objectives are to determine the adverse outcomes of hypothermia and warming measures

DETAILED DESCRIPTION:
Background Hypothermia, defined as core body temperature less than 36 degrees Celsius, occurs frequently during the course of surgery in patients across all ages, especially in the young. It causes significant medical consequences including cardiac events, bleeding, surgical site infection, increased shivering and patient discomfort, as well as longer hospital stays. Although guidelines exist for health care providers in terms of temperature management during surgery, these guidelines are not always followed as the warming measures can be costly, for example, single-use temperature probes and disposable blankets, with potential risks of the equipment overheating causing burns and contamination during surgery

Methodology The investigators aim to include up to 6,000 children presenting for either scheduled or emergency surgeries. Core temperature before, during and after surgery using routine temperature monitoring devices such as tympanic, axillary, oral, rectal and SPOTON (a non-invasive method using a sticker placed on the forehead) will be measured. Other outcomes collected will include cardiac arrhythmias, blood loss, hyperthermia, burn injuries, shivering, discomfort, length of PACU and length of hospitalization, wound infection rates, . Patients will receive the usual heat-loss prevention and warming measures.

Interim analysis of the first 2000 patients using the SPOTON method of continuous core temperature monitoring will be done to determine incidence and duration of peri-operative hypothermia. This monitoring modality will be compared for agreement with the conventional tympanic and forehead infra-red thermoscan methods. Patient and perioperative risk factors predisposing to hypothermia will be identified to guide in the formulation of clinical practice guidelines tailored to the local population. Guidelines will be implemented, and post-implementation incidence of IPH will be determined A pre- versus post-implementation cost analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric patients ages 16 and younger undergoing elective or emergency surgeries in paediatric major and day surgical operating theaters in KK women's and Children's Hospital.

Exclusion Criteria:

* Patients undergoing operative procedures under local anaesthesia
* Patients with impaired temperature control e.g., severe head injury, febrile illness
* Patients who are admitted to intensive care unit (ICU) post-operatively.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruitment of participants: consecutive sampling of eligible participants recruited from daily operating lists in major and day surgery operating theatres
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence (%) of perioperative hypothermia | From induction of anaesthesia to discharge from PACU, approximately 8 hours
  Hypothermia is defined as Core temperature<36 degrees Celsius. Incidence of hypothermia is the occurence of hypothermia, measured in percentage(%).
Duration (minutes) of perioperative hypothermia | From induction of anaesthesia to discharge from PACU, approximately 8 hours
  Hypothermia is defined as Core temperature<36 degrees Celsius. Duration of hypothermia is defined as the duration of time in minutes where temperature is less than 36 degrees celsius.

SECONDARY OUTCOMES:
Incidence of short term adverse outcomes of IPH in the paediatric population | From induction of anaesthesia to discharge from PACU, approximately 8 hours
  Short term adverse outcomes include intra-operative blood loss, arrhythmia, post-anaesthesia shivering, discomfort from cold, PACU stay
Incidence of long term adverse outcomes of IPH in the paediatric population | From PACU discharge time up to 6 months post-surgery
  Long term outcomes include: surgical site infection and hospitalization stay
Incidence of adverse outcomes of warming interventions in the paediatric population eg. Hyperthermia and burns injury | From induction of anaesthesia to discharge from PACU, approximately 8 hours
  Hyperthermia cTemp >38 ºC, burns injury

CONTACTS AND LOCATIONS:
Overall Officials: Shu Ying Lee, FANZCA, Mmed, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided